CLINICAL TRIAL: NCT06915740
Title: Virtual Pulmonary Rehabilitation Program for COPD Patients; a Pilot Study
Acronym: e-PURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Matthijs Feuth, MD PhD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1649/2024
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: copd; pulmonary rehabilitation; telemedicine; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual pulmonary rehabilitation (Other): Participation in a virtual pulmonary rehabilitation program developed by a multidisciplinary team
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — virtual rehabilitation, including endurance exercise, strength training, breathing exercises, patient education, dietary advice

SUMMARY:
The goal of this pilot study is to investigate the feasibility of a virtual rehabilitation program in COPD patients. The main questions it aims to answer are:

1. To facilitate a safe rollout of the remote rehabilitation program for COPD patients in Southwest Finland.
2. To identify and subsequently improve limitations of the rehabilitation program.
3. To evaluate the levels of participant engagement and adherence to the digital COPD rehabilitation program over an extended period to understand its sustainability and long-term impact.
4. To determine the effectiveness of the digital COPD rehabilitation program in improving lung function, exercise capacity, and quality of life among participants
5. To assess the impact of the digital program on healthcare resource utilization, including hospital readmissions, emergency room visits, and outpatient visits related to COPD management.
6. To measure participant satisfaction, usability, and overall experience with the digital platform to identify areas for improvement and enhance user engagement.
7. To evaluate the cost-effectiveness of implementing the digital program compared to conventional rehabilitation methods, considering direct healthcare costs.

Participants will be enrolled in a virtual rehabilitation program, and a proportion of the patients is invited for focus group discussion to assess their experiences.

DETAILED DESCRIPTION:
The e-PURE study is an investigator initiated study, which aims to evaluate the feasibility, effectiveness, and long-term outcomes of a digital pulmonary rehabilitation program designed for patients with Chronic Obstructive Pulmonary Disease (COPD) in Southwest Finland. This pilot study assesses patient adherence, lung function, exercise capacity, quality of life, and the program's potential impact on healthcare utilization.

COPD is a common disease, affecting mostly elderly, with significant impact on life expectancy and quality of life. Pulmonary rehabilitation (PR) is an essential intervention for COPD patients, known to enhance health-related quality of life and reduce symptoms like shortness of breath. Traditional PR programs are underutilized due to accessibility barriers, with less than 1% of COPD patients in Canada and 3.7% in the U.S. attending such programs. The COVID-19 pandemic exacerbated these challenges by halting in-person PR programs. Virtual PR offers a promising, non-inferior alternative. The e-PURE study responds to this need by rolling out a digital rehabilitation program developed by a multidisciplinary team of healthcare professionals.

This is a single-arm observational pilot study enrolling up to 50 COPD patients. The rehabilitation program spans around 12 weeks, with follow-up assessments at 16 and 26 weeks post-enrolment. Patients undergo a tailored rehabilitation plan that includes individualized exercise routines, nutritional counselling, and smoking cessation support. Progress is reported through questionnaires and clinical evaluations such as the 6-minute walk test.

The primary outcome measure is the improvement in distance during the 6-minute walk test after the program, compared to baseline. Secondary outcomes include patient satisfaction, changes in the St. George Respiratory Questionnaire, and healthcare resource utilization (hospital readmissions, emergency visits).

The pilot study will identify whether a larger follow-up study is feasible, and indicate the number of patients to recruit.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the remote rehabilitation program for COPD patients, fulfilling criteria 1a, 1b and 1c 1a Documented COPD diagnosis (ICD 10 code J44) 1b Expected survival > 1 year 1c Sufficient technical and language skills for safe participation in the program
2. Signed informed consent

Exclusion Criteria:

* Severe comorbidities with expected survival of less than 1 year
* Clinical suspicion that remote rehabilitation may be unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking test | from enrollment to 16-26 weeks
  6 minutes walking test after the rehabilitation program in comparison to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Turku University Hospital, Turku, Southwest Finland
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No
Privacy policy does not allow to share individual participant data

REFERENCES:
- [Background] Holland AE, Cox NS, Houchen-Wolloff L, Rochester CL, Garvey C, ZuWallack R, Nici L, Limberg T, Lareau SC, Yawn BP, Galwicki M, Troosters T, Steiner M, Casaburi R, Clini E, Goldstein RS, Singh SJ. Defining Modern Pulmonary Rehabilitation. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2021 May;18(5):e12-e29. doi: 10.1513/AnnalsATS.202102-146ST. PMID 33929307
- [Background] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Background] Janjua S, Banchoff E, Threapleton CJ, Prigmore S, Fletcher J, Disler RT. Digital interventions for the management of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD013246. doi: 10.1002/14651858.CD013246.pub2. PMID 33871065

DOCUMENTS (1):
  • Study Protocol (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT06915740/Prot_000.pdf